CLINICAL TRIAL: NCT04373681
Title: Validity and Reliability of the Turkish Version of Western Ontario Osteoarthritis of the Shoulder Index
Brief Title: Validity and Reliability of the Turkish Version of WOOS
Status: Completed | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Şeyda ÖZAL, Research Asistant, Gazi University
Other Study IDs: Gazi Unv
Record Dates: First submitted 2020-04-27; First posted 2020-05-04 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Evaluating the Validity and Reliability of the Turkish WOOS
Keywords: WOOS; validation; Osteoarthritis; Shoulder; Turkish; Version
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: patient-administered questionnaires — patient-administered questionnaires

SUMMARY:
Various clinical scales are available to investigate shoulder diseases. Some of them, culturally adapted to the Turkish population. However, none of them are specific for osteoarthritis of the shoulder. Thus, this study aimed to translate the WOOS index into Turkish and investigate its psychometric properties in the Turkish population.

DETAILED DESCRIPTION:
Purpose; The aim of this study is to adapt the Western Ontario Osteoarthritis of the Shoulder Index (WOOS) specific to shoulder osteoarthritis, to Turkish and evaluate its validity and reliability.

Methods; WOOS index was translated and culturally adapted to Turkish, systematically. It was applied to 68 patients with osteoarthritis of the shoulder treated conservatively. The reliability of the scale was checked through internal consistency and test-retest methods. Internal consistency was analyzed with Cronbach's alpha value. Test-retest reliability was assessed using an intraclass correlation coefficient with 25 patients. The Western Ontario Rotator Cuff (WORC), The Shoulder Pain and Disability Index (SPADI), and The Society of American Shoulder and Elbow Surgeons Standardized Shoulder Assessment (ASES) score were used to conduct concurrent validity.

ELIGIBILITY:
Inclusion Criteria:

* Presence of the shoulder osteoarthritis, to be a native Turkish speaker

Exclusion Criteria:

* Illiteracy, cognitive impairment, presence of shoulder circumference fractures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult male and female patients with osteoarthritis of the shoulder
Sampling Method: Non-Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2017-12-04 (Actual); Primary Completion 2020-01-10 (Actual); Study Completion 2020-03-15 (Actual)

PRIMARY OUTCOMES:
Western Ontario Osteoarthritis of the Shoulder Index, patients get a minimum of 0 points (best condition) and a maximum of 1900 points (worst condition) on this scale. | 1st day
  patient administered, spesific to osteoarthritis of shoulder, multisectional questionnaire
Western Ontario Osteoarthritis of the Shoulder Index, patients get a minimum of 0 points (best condition) and a maximum of 1900 points (worst condition) on this scale. | 2 days later
  patient administered, spesific to osteoarthritis of shoulder, multisectional questionnaire
The Western Ontario Rotator Cuff Index, patients get a minimum of 0 points (best condition) and a maximum of 2100 points (worst condition) on this scale. | 1st day
  patient administered, spesific to rotator cuff disease, multisectional questionnaire
The Shoulder Pain and Disability Index, patients get a minimum of 0 points (best condition) and a maximum of 100 points (worst condition) on this scale. | 1st day
  patient administered, spesific to upper limp, two sectional questionnaire
The Society of American Shoulder and Elbow Surgeons Standardized Shoulder Assessment, patients get a minimum of 0 points (worst condition) and a maximum of 100 points (best condition) on this scale. | 1st day
  patient administered, spesific to upper limp, two sectional questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Nevin A GÜZEL, Prof, Principal Investigator — Gazi University Faculty of Health Sciences; Şeyda ÖZAL, MSc, Study Chair — Gazi University Faculty of Health Sciences; Ahmet Y KAPTAN, MD, Study Chair — Dr. Sami Ulus Hospital; Nihan KAFA, Assc Prof, Study Chair — Gazi University Faculty of Health Sciences; Toygun K EREN, MD, Study Chair — Ankara Training and Research Hospital
Locations (3):
- Turkey (Türkiye) (3):
  - Dr. Sami Ulus Maternity, Child Health and Diseases Training and Research Hospital, Department of Orthopaedics & Traumatology, Ankara
  - Ankara Training and Research Hospital, Department of Orthopaedics & Traumatology, Ankara
  - Gazi University Faculty of Health Sciences Physiotherapy and Rehabilitation Department, Ankara

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Petersson CJ. Degeneration of the gleno-humeral joint. An anatomical study. Acta Orthop Scand. 1983 Apr;54(2):277-83. doi: 10.3109/17453678308996570. PMID 6846007
- [Background] Ozer M, Ataoglu MB, Cetinkaya M, Ayanoglu T, Kaptan AY, Kanatli U. Do intra-articular pathologies accompanying symptomatic acromioclavicular joint degeneration vary across age groups? Eklem Hastalik Cerrahisi. 2019 Apr;30(1):2-9. doi: 10.5606/ehc.2019.62431. PMID 30885102
- [Background] Millett PJ, Gobezie R, Boykin RE. Shoulder osteoarthritis: diagnosis and management. Am Fam Physician. 2008 Sep 1;78(5):605-11. PMID 18788237
- [Background] Lo IK, Griffin S, Kirkley A. The development of a disease-specific quality of life measurement tool for osteoarthritis of the shoulder: The Western Ontario Osteoarthritis of the Shoulder (WOOS) index. Osteoarthritis Cartilage. 2001 Nov;9(8):771-8. doi: 10.1053/joca.2001.0474. PMID 11795997
- [Background] Tugay U, Tugay N, Gelecek N, Ozkan M. Oxford Shoulder Score: cross-cultural adaptation and validation of the Turkish version. Arch Orthop Trauma Surg. 2011 May;131(5):687-94. doi: 10.1007/s00402-010-1242-9. Epub 2010 Dec 30. PMID 21191606
- [Background] Celik D, Atalar AC, Demirhan M, Dirican A. Translation, cultural adaptation, validity and reliability of the Turkish ASES questionnaire. Knee Surg Sports Traumatol Arthrosc. 2013 Sep;21(9):2184-9. doi: 10.1007/s00167-012-2183-3. Epub 2012 Aug 30. PMID 22932692
- [Background] Najafov E, Ozal S, Kaptan AY, Ulucakoy C, Kanatli U, Ataoglu B, Basar S. Validity and Reliability of the Turkish Version of LHB Score. J Sport Rehabil. 2020 Mar 4;30(1):30-36. doi: 10.1123/jsr.2019-0364. PMID 32131050
- [Background] Celik D. Turkish version of the modified Constant-Murley score and standardized test protocol: reliability and validity. Acta Orthop Traumatol Turc. 2016;50(1):69-75. doi: 10.3944/AOTT.2016.14.0354. PMID 26854052
- [Background] Beaton D, Bombardier C, Guillemin F, Ferraz MB (2002) Recommendations for the cross-cultural adaptation of health status measures. New York: American Academy of Orthopaedic Surgeons 12:1-9
- [Background] El O, Bircan C, Gulbahar S, Demiral Y, Sahin E, Baydar M, Kizil R, Griffin S, Akalin E. The reliability and validity of the Turkish version of the Western Ontario Rotator Cuff Index. Rheumatol Int. 2006 Oct;26(12):1101-8. doi: 10.1007/s00296-006-0151-2. Epub 2006 Jun 24. PMID 16799776
- [Background] Bumin G, Tüzün EH, Tonga E (2008) The Shoulder Pain and Disability Index (SPADI): Cross-cultural adaptation, reliability, and validity of the Turkish version. Journal of Back and Musculoskeletal Rehabilitation 21(1):57-62
- [Background] Snyder CF, Aaronson NK, Choucair AK, Elliott TE, Greenhalgh J, Halyard MY, Hess R, Miller DM, Reeve BB, Santana M. Implementing patient-reported outcomes assessment in clinical practice: a review of the options and considerations. Qual Life Res. 2012 Oct;21(8):1305-14. doi: 10.1007/s11136-011-0054-x. Epub 2011 Nov 3. PMID 22048932
- [Background] Weir JP. Quantifying test-retest reliability using the intraclass correlation coefficient and the SEM. J Strength Cond Res. 2005 Feb;19(1):231-40. doi: 10.1519/15184.1. PMID 15705040
- [Background] Klintberg IH, Lind K, Marlow T, Svantesson U. Western Ontario Osteoarthritis Shoulder (WOOS) index: a cross-cultural adaptation into Swedish, including evaluation of reliability, validity, and responsiveness in patients with subacromial pain. J Shoulder Elbow Surg. 2012 Dec;21(12):1698-705. doi: 10.1016/j.jse.2011.11.027. Epub 2012 Mar 21. PMID 22445627
- [Background] Rasmussen JV, Jakobsen J, Olsen BS, Brorson S. Translation and validation of the Western Ontario Osteoarthritis of the Shoulder (WOOS) index - the Danish version. Patient Relat Outcome Meas. 2013 Sep 18;4:49-54. doi: 10.2147/PROM.S50976. eCollection 2013. PMID 24133377
- [Background] Corona K, Cerciello S, Morris BJ, Visona E, Merolla G, Porcellini G. Cross-cultural adaptation and validation of the Italian version of the Western Ontario Osteoarthritis of the Shoulder index (WOOS). J Orthop Traumatol. 2016 Dec;17(4):309-313. doi: 10.1007/s10195-016-0400-4. Epub 2016 Mar 31. PMID 27033229
- [Background] Jia ZY, Zhang C, Cui J, Xue CC, Xu WD. Translation and validation of the Simplified Chinese version of Western Ontario Osteoarthritis of the Shoulder Index (WOOS). Medicine (Baltimore). 2018 Mar;97(13):e8691. doi: 10.1097/MD.0000000000008691. PMID 29595694